CLINICAL TRIAL: NCT06297798
Title: Effects of Telerehabilitation-Based Interventions on the Musculoskeletal System in Drivers: A Crossover Longitudinal Study
Brief Title: Effects of Telerehabilitation-Based Interventions on the Musculoskeletal System in Drivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya Applied Sciences University (Other)
Responsible Party: Principal Investigator, Pakize Nurgul Sen, Research Assistant, Sakarya Applied Sciences University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SakaryaAppliedSciencesUPNS
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Drive; Musculoskeletal Diseases; Postural; Defect
Keywords: drivers, musculoskeletal system disease, posture, longitudinal study
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): In the telerehabilitation group, posture and stabilization exercises will be performed using Whatsapp and Zoom applications for 40 minutes, 5 days a week. Exercises will be applied for 10 weeks.
  Posture and Stabilization Exercise Program:
  1. Stretching of neck flexor, extensor, and lateral flexor muscles (30 seconds each)
  2. Pectoral muscle stretching (30 seconds, 3 repetitions)
  3. Isometric neck exercises (10 seconds, 10 repetitions)
  4. Rhomboid strengthening exercise (bringing shoulder blades closer together against resistance using a TheraBand) (10 seconds, 10 repetitions)
  5. Stretching of hamstring, lumbar lordosis and gastrocnemius muscles (sitting and standing) (30 seconds, 3 repetitions)
  6. Pelvic posterior tilt exercise (10 seconds, 10 repetitions)
  7. Bridge exercise (20 seconds, 10 repetitions)
  8. Single-leg bridge exercise (Right-Left) (10 seconds, 10 repetitions)
  9. Plank (starting with 60 seconds, increasing by 10 seconds each week)
  Interventions: Other: Telerehabilitation
- Control Group (No Intervention): The control group will not be given any exercise program; instead, general posture recommendations will be given.

INTERVENTIONS:
Other: Telerehabilitation — The telerehabilitation program will be implemented using Whatsapp and Zoom applications for 40 minutes, 5 days a week. Posture and stabilization exercises will be performed, and the exercises will be performed for 10 weeks.
  Posture and Stabilization Exercise Program:
  1. Stretching of neck flexor, extensor, and lateral flexor muscles (30 seconds each)
  2. Pectoral muscle stretching (30 seconds, 3 repetitions)
  3. Isometric neck exercises (10 seconds, 10 repetitions)
  4. Rhomboid strengthening exercise (bringing shoulder blades closer together against resistance using a TheraBand) (10 seconds, 10 repetitions)
  5. Stretching of hamstring, lumbar lordosis and gastrocnemius muscles (sitting and standing) (30 seconds, 3 repetitions)
  6. Pelvic posterior tilt exercise (10 seconds, 10 repetitions)
  7. Bridge exercise (20 seconds, 10 repetitions)
  8. Single-leg bridge exercise (Right-Left) (10 seconds, 10 repetitions)
  9. Plank (starting with 60 seconds, increasing by 10 seconds each week)
  Arms: Telerehabilitation Group

SUMMARY:
This study is designed to examine the effect of telerehabilitation application on the musculoskeletal system of drivers.The study will include 40 voluntary participants who work as drivers on inter-district routes in Sakarya. The participants' sociodemographic information, musculoskeletal problems, and postures will be assessed. Participants will be divided into two groups: one group will receive tele-rehabilitation with posture and stabilization exercises, while the other group will serve as the control group. The exercises will be implemented for 10 weeks, followed by an 8-week tapering period, after which the groups will be crossed over. A re-evaluation will be conducted after 10 weeks, with follow-up assessments scheduled for 3 months later.

DETAILED DESCRIPTION:
The aim of the research is to investigate the effectiveness of telerehabilitation-based interventions in the management and improvement of common musculoskeletal disorders prevalent among drivers. This study will longitudinally examine the potential effects of developing and implementing customized posture and stabilization exercise programs for reducing posture and musculoskeletal disorders in drivers. The goal is to provide evidence of the effectiveness of telerehabilitation applications on the musculoskeletal health of drivers.

The study plans to involve 40 male volunteers aged 30-65 engaged in inter-district driving in Sakarya. Inclusion criteria for the study include working as an inter-district driver, driving a vehicle for at least 6 hours per day for a minimum of one year, and the ability to use at least one of the WhatsApp, Zoom, or Teams applications. Exclusion criteria include undergoing orthopedic surgery in the past year and a lack of consent to participate in the study. Within the scope of the study, sociodemographic information will be collected from all participants, their postures will be assessed using the "posture screen" application, and musculoskeletal problems will be evaluated using the "Cornell Musculoskeletal Disorders Questionnaire."

At the end of the assessment, participants will be divided into two groups using the layered randomization method. The intervention group will receive posture and stabilization exercises through telerehabilitation via WhatsApp, Zoom, or Teams applications for 45 minutes per day, five days a week, for 10 weeks. General advice will be given to both groups, but no exercise program will be provided to the control group. After 10 weeks, the same assessments will be conducted for both the control and intervention groups. Subsequently, an 8-week tapering period will be expected, followed by the crossover of the groups. Those initially in the intervention group will form the control group, and vice versa.

After 10 weeks of training, the same assessments will be conducted again, and following this assessment, a final evaluation will be conducted 3 months later to complete the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals working as drivers in intercity minibuses in Sakarya.
* Those who have been working as drivers for at least one year.
* Age between 30 and 65.
* Male gender.
* Those who can use a smartphone.
* Those who can use at least one of the following applications: WhatsApp, Zoom, or Teams.

Exclusion Criteria:

* Orthopedic surgeries undergone within the past year.
* Inability to obtain consent to participate in the study.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will be conducted only on male drivers.
Enrollment: 40 (Estimated)
Dates: Start 2024-03-14 (Estimated); Primary Completion 2024-03-21 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
MUSCLE SKELETAL SYSTEM ASSESSMENT | Through study completion, an average of 1 year
  The Cornell Musculoskeletal System Questionnaire will be used for musculoskeletal system evaluation. While conducting the survey, the illnesses experienced by the employees in the last week are taken as basis. In this survey, neck, shoulder (right-left), back, upper arm (right-left), waist, forearm (right-left), wrist (right-left), hip, upper leg (right-left), knee. Questions are asked for 20 body parts such as (right-left), lower leg (right-left) and foot (right-left) and the risk score is calculated as a result of the answers received. While calculating the relevant score, risk scores are calculated separately for each body region by multiplying scores such as the number of times the employee has experienced the discomfort in the current area, the severity of the discomfort felt and the obstacle in working. The final total score is calculated. A high score indicates high discomfort.

SECONDARY OUTCOMES:
Posture Measures | Through study completion, an average of 1 year
  Posture evaluation will be made using the "PostureScreen Mobile" application. This application is a reliable and valid mobile tool designed specifically to assess static posture and, in particular, forward head tilt. All participants will be allowed to wear thin, tight clothing provided that reference anatomical landmarks are clearly visible. All evaluations will be repeated in the same place and under the same conditions. The photo will always be taken from a distance of 10 feet (approximately 3.5 meters) and from a height of 3.5 feet (approximately 1.5 meters).

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University of Applied Sciences, Sakarya, Turkey (Türkiye)